CLINICAL TRIAL: NCT01467635
Title: Endobronchial Ultrasound Transbronchial Needle Aspiration (EBUS-TBNA) Versus Endobronchial Ultrasound Transbronchial Needle Biopsy (EBUS-TBNB) in the Assessment of Mediastinal and Hilar Lymphadenopathy: a Randomised Trial
Brief Title: EBUS-TBNA Versus EBUS-TBNB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Manufacturer did not develop and deliver the necessary biopsy forceps needles in time
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other); Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2011PA002B
Record Dates: First submitted 2011-11-04; First posted 2011-11-09 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Mediastinal Lymphadenopathy; Hilar Lymphadenopathy; Carcinoma; Lymphoma; Sarcoidosis; Mycobacterial Disease
Keywords: Endobronchial ultrasound; Transbronchial needle aspiration; Transbronchial biopsy forceps; Mediastinal lymphadenopathy; Hilar lymphadenopathy
MeSH Terms: conditions — Carcinoma; Lymphoma; Sarcoidosis; Mycobacterium Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBUS-TBNA (Active Comparator): Sampling using endobronchial ultrasound guided transbronchial needle aspiration
  Interventions: Device: Endobronchial ultrasound guided lymph node sampling
- EBUS-TBNB (Experimental): Sampling using endobronchial ultrasound guided transbronchial forceps biopsy needle.
  Interventions: Device: Endobronchial ultrasound guided lymph node sampling

INTERVENTIONS:
Device: Endobronchial ultrasound guided lymph node sampling — Patients with enlarged mediastinal or hilar lymph nodes have these sampled under endobronchial ultrasound guidance using either the EBUS-TBNA needle or the EBUS-TBNB biopsy forceps.
  Other Names: Olympus EBUS-TBNA needle; Olympus EBUS-TBNB biopsy forceps

SUMMARY:
A prospective diagnostic clinical study randomising patients undergoing endobronchial ultrasound guided transbronchial needle aspiration (EBUS-TBNA) of enlarged mediastinal and hilar lymph nodes to have sampling using the usual EBUS-TBNA needle or a novel biopsy forceps (EBUS-TBNB).

The study aims to establish whether the use of EBUS-TBNB can significantly increase the diagnostic yield over EBUS-TBNA, without an increase in complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for EBUS-TBNA as part of clinical care
* Lymph nodes larger than 10mm in diameter
* Age > 18 years
* Able to provide written informed consent

Exclusion Criteria:

* Contraindications for needle or forceps biopsy (e.g. coagulopathy, anticoagulation, thrombocytopenia)
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The percentage of lymph nodes sampled resulting in a definitive diagnosis (as defined in the protocol) in the two study arms. | 18 months
  The definition of a "definitive diagnosis" is dependant on the diagnosis and is clarified below:
  * Carcinoma/lymphoma: The lymph node sample is adequate to make a diagnosis as well as provide immunohistochemistry information enabling subtyping of the tumour.
  * Sarcoidosis: The presence of well formed epithelioid non-caseating granulomas.
  * Mycobacterial infection: The presence of caseating granulomas, positive Ziehl Nielson staining for acid fast bacilli, or the tissue successfully cultures Mycobacterium.

SECONDARY OUTCOMES:
The difference in the complication rate between the two study arms | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Zoumot, MBBS, MRCP, MSc, Study Director — Royal Brompton Hospital NHS Foundation Trust, Chelsea and Westminster Hospital NHS Fundation Trust; Pallav L Shah, MD, FRCP, Principal Investigator — Royal Brompton Hospital NHS Foundation Trust, Chelsea and Westminster Hospital NHS Foundation Trust
Locations (3):
- Thoraxklinik, University of Heidelberg, Heidelberg, Germany
- United Kingdom (2):
  - Chelsea and Westminster Hospital, London
  - The Royal Brompton Hospital, London